CLINICAL TRIAL: NCT02420366
Title: Multi-center, Retrospective Study of Cases of Serious Infections Due to Carbapenem-Resistant Enterobacteriaceae
Brief Title: Study of Cases of Serious Infections Due to Carbapenem-Resistant Enterobacteriaceae
Status: Completed | Type: Observational
Sponsor: Rempex (a wholly owned subsidiary of Melinta Therapeutics, Inc.) (Industry)
Responsible Party: Sponsor
Organization: Melinta Therapeutics, Inc. (Industry)
Other Study IDs: Rempex 506 NH
Record Dates: First submitted 2015-04-08; First posted 2015-04-17 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Urinary Tract Infection, Complicated; Acute Pyelonephritis; Hospital Acquired Bacterial Pneumonia; Ventilator-associated Bacterial Pneumonia; Bacteremia
MeSH Terms: conditions — Urinary Tract Infections; Bacteremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A multi-center, retrospective study of cases of serious bacterial infections including complicated Urinary Tract Infection (cUTI) or Acute Pyelonephritis (AP), Hospital Acquired Bacterial Pneumonia (HABP), Ventilator Acquired Bacterial Pneumonia (VABP), and/or bacteremia caused by Carbapenem-Resistant Enterobacteriaceae (CRE)

DETAILED DESCRIPTION:
This multi-center, retrospective study of cases of serious bacterial infections (including cUTI or AP, HABP, VABP, and/or bacteremia caused by CRE) will consist of a chart review over a 6 month period from September 1, 2013 to March 1, 2014. De-identified data will be collected from the chart review of at least 150 cases of selected infections due to CRE at approximately 20 sites.

The study itself is strictly observational and retrospective, with no direct study-related patient interaction, treatment, or testing. There will be no patient identifying data collected as part of this study.

Charts of patients who meet study-defined criteria for cUTI or AP, HABP, VABP, and/or bacteremia and have a culture from the site of infection or the blood that is positive for a Carbapenem-Resistant Enterobacteriaceae will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age.
* Carbapenem resistant Enterobacteriaceae (CRE) must be identified in the urine, blood or respiratory tract samples submitted for culture in the setting of cUTI or AP, HABP, VABP, and/or bacteremia.
* Diagnosis with either cUTI or AP, HABP, VABP, and/or bacteremia.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with serious CRE infections identified by chart review at up to 20 sites
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of positive CRE infections (specifically cUTI, AP, HABP, VABP, Bacteremia) in a target patient population | 6 month period from September 1, 2013 to March 1, 2014

CONTACTS AND LOCATIONS:
Overall Officials: Karen Fusaro, Study Director — Sponsor GmbH
Locations (20):
- United States (11):
  - Chicago, Illinois
  - Evanston, Illinois
  - Detroit, Michigan
  - New Brunswick, New Jersey
  - Somers Point, New Jersey
  - New York, New York
  - Rochester, New York
  - Durham, North Carolina
  - Cleveland, Ohio
  - Pittsburgh, Pennsylvania
  - Charlottesville, Virginia
- Athens, Greece
- Italy (7):
  - Bologna
  - Florence
  - Genova
  - Pisa
  - Roma
  - Rome
  - Udine
- Manchester, United Kingdom